CLINICAL TRIAL: NCT00525161
Title: A Phase II Study of Adding the Multikinase Inhibitor Sorafenib (Nexavar) to Existing Endocrine Therapy in Patients With Advanced Breast Cancer
Brief Title: Study Adding Multikinase Inhibitor Sorafenib to Existing Endocrine Therapy in Patients With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and loss of funding
Sponsor: Suleiman Massarweh (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Suleiman Massarweh, Clinical Faculty, Internal Medicine / Oncology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-BRE-41-BP
Record Dates: First submitted 2007-09-03; First posted 2007-09-05 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; Sorafenib; Nexavar; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib & Endocrine Therapy (Experimental): Sorafenib & Endocrine Therapy
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — 400 mg PO (orally) twice daily for 12 months from study enrollment or until disease progression, whichever occurs first.
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to determine the clinical response rate to sorafenib when added to existing endocrine therapy in patients with advanced breast cancer.

DETAILED DESCRIPTION:
A pilot Phase II study adding sorafenib to endocrine therapy in 11 patients with metastatic estrogen receptor-positive breast cancer was conducted. Primary end point was response by Response Evaluation Criteria in Solid Tumors (RECIST) after 3 months of sorafenib. Secondary end points included safety, time to progression and biomarker modulation. The study closed early owing to slow accrual.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be female.
* Age ≥ 18 years old.
* Histologically proven carcinoma of the breast.
* Estrogen receptor and/or Progesterone positive disease.
* Metastatic or locally advanced disease.
* Patients on a preexisting endocrine agent for at least 3 months before enrollment.
* Have residual measurable disease after

  1. maximal response to endocrine therapy or
  2. no response to endocrine therapy or
  3. progressive non-visceral disease on endocrine therapy.
* Must be able to provide a tumor block from either the primary or metastatic site, if available.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Adequate organ function.

Exclusion Criteria:

* Patients with rapidly progressive disease on endocrine therapy who would otherwise be candidates for chemotherapy.
* Other coexisting malignancies, with the exception of basal cell carcinoma or cervical carcinoma in situ.
* Prior use of anti-angiogenic agents.
* As judged by the investigator, uncontrolled intercurrent illness.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* A serious non-healing wound or ulcer.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within the 4 weeks prior to the first dose of the study drug.
* Pulmonary hemorrhage/bleeding event ≥ Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2 within the 4 weeks prior to the first dose of study drug.
* Pregnancy
* Any condition that impairs patient's ability to swallow whole pills.
* Documented malabsorption problem.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-10; Primary Completion 2013-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suleiman Massarweh, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Result] Massarweh S, Moss J, Wang C, Romond E, Slone S, Weiss H, Karabakhtsian RG, Napier D, Black EP. Impact of adding the multikinase inhibitor sorafenib to endocrine therapy in metastatic estrogen receptor-positive breast cancer. Future Oncol. 2014 Dec;10(15):2435-48. doi: 10.2217/fon.14.99. PMID 24826798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were recruited from the University of Kentucky Markey Cancer Center from November 2009-November 2011.
Period: Overall Study
Arm/Group | Sorafenib & Endocrine Therapy
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib & Endocrine Therapy
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 45 [39 to 72]
Age, Customized [Number; unit: participants]
  <40 years | 3
  40-49 years | 3
  50-59 years | 1
  60-69 years | 2
  >=70 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Locally advanced [Number; unit: participants]
  Yes | 5
  No | 6
Relapsed versus de novo metastasis [Number; unit: participants]
  de novo | 7
  Relapsed | 4
Estrogen receptor status [Number; unit: participants]
  Positive | 11
  Negative | 0
Progesterone receptor status [Number; unit: participants]
  Positive | 9
  Negative | 2
Human epidermal growth factor receptor 2 (HER2) status [Number; unit: participants]
  Negative | 9
  Unknown | 2
Endocrine therapy at study entry [Number; unit: participants]
  Tamoxifen | 7
  Anastrozole | 1
  Exemestane | 1
  Fulvestrant | 1
  Letrozole | 1
Line of current endocrine therapy [Number; unit: participants]
  First-line (Primary) treatment | 9
  Second-line (Subsequent) treatment | 2
Disease status at entry [Number; unit: participants]
  Progressive Disease | 8
  Stable disease with maximal response | 3
Prior chemotherapy [Number; unit: participants]
  No | 8
  Yes | 3
Bone metastases [Number; unit: participants]
  Yes | 9
  No | 2
Lung Metastases [Number; unit: participants]
  Yes | 5
  No | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Patients were followed monthly for clinical and toxicity evaluation. Disease response by RECIST criteria v1.0 was assessed after 3 months by appropriate scans and these were obtained every 2 months thereafter until progression.
Time Frame: 12 weeks after treatment & 8 weeks after initial documentation of response
Population: one discontinued treatment after 2 weeks owing to a grade 3 rash and was not evaluable for response
Measure: Number; unit: participants
Arm/Group | Sorafenib & Endocrine Therapy
Number analyzed (Participants) | 10
participants
  Stable Disease | 7
  Progression | 3
Statistical Analysis 1: Comparison: Sorafenib & Endocrine Therapy; Based on known historical response rate to sorafenib of no better than 5-10%, the study was designed to test the null hypothesis that the clinical response rate is no better than 10% versus the alternative hypothesis that it is at least 25% when sorafenib is added to endocrine therapy. In the first stage, 18 patients were planned for enrollment, and if two or fewer responses were observed, the trial would be terminated. The study stopped after 11 due to slow accrual and withdrawal of funding; Test type: Superiority or Other; Clinical Response Rate at 3 months = 0 — Defined as complete response/partial response after 3 months of adding sorafenib to endocrine therapy

2. Secondary Outcome: Time to Progression
Time Frame: continuously
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib & Endocrine Therapy
Number analyzed (Participants) | 11
months | 6.1 [2.6 to 11.3]
Statistical Analysis 1: Comparison: Sorafenib & Endocrine Therapy; Test type: Superiority or Other; Median Progression Free Survival = 6.1, 95% CI 2-sided [2.6 to 11.3]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as complete response, partial response, or stable disease (CR/PR/SD) as measured by Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for a minimum of at least 24 weeks.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib & Endocrine Therapy
Number analyzed (Participants) | 10
percentage of participants | 50 [19 to 81]

ADVERSE EVENTS:
Arm/Group | Sorafenib & Endocrine Therapy
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib & Endocrine Therapy (N=11)
Infection/Herpes Zoster (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib & Endocrine Therapy (N=11)
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 9
Weight Loss (Investigations) | 9
Hypertension (Vascular disorders) | 6
Nausea/vomiting (Gastrointestinal disorders) | 6
Elevated ALT/AST (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Fatigue (General disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination of study due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No